CLINICAL TRIAL: NCT05610033
Title: Pilot evaluatIon Of NovEl tEmpoRary ExtraVascular PACING (PIONEER EV PACING) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AtaCor Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DOC-10219
Record Dates: First submitted 2022-10-30; First posted 2022-11-08 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Conduction Defect
Keywords: Temporary Ventricular Pacing; Extravascular
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AtaCor EV Temporary Pacing Lead System (Experimental): Subjects implanted with the AtaCor StealthTrac Lead Model AC-101400
  Interventions: Device: AtaCor StealthTrac Lead

INTERVENTIONS:
Device: AtaCor StealthTrac Lead — Subjects will receive the AtaCor StealthTrac Lead being evaluated in the study.

SUMMARY:
The PIONEER EV PACING Study is prospective, multi-center, acute (in-hospital), single-arm, pilot study. The study objective is to characterize preliminary safety and performance of the AtaCor EV Temporary Pacing Lead System when used as intended for clinical use as a temporary pacing lead.

DETAILED DESCRIPTION:
The primary safety endpoint is freedom from Adverse Device Effects, CTCAE Grade 3 or higher. The primary performance endpoint is percentage of Subjects with demonstrated pacing capture following lead fixation.

Up to 30 subjects will be enrolled at up to three (3) investigation centers. Enrolled subjects will undergo insertion of a StealthTrac Lead within one calendar day of an eligible planned index procedure that requires a temporary pacing lead. Echocardiographic evaluations will be performed before and after StealthTrac Lead insertion, as well as after the index procedure, to assess for pericardial effusion. Post-operative fluoroscopic images are required in all subjects to document the final lead position. In subjects without an underlying ventricular escape rhythm, a concomitant, commercially available pacing lead is required. Lead measurements (Thresholds, Impedance, R-Waves) and an insertion procedure survey will be obtained.

Subjects will be restricted to bed rest while the StealthTrac lead remains inserted. The StealthTrac Lead will be connected to a commercially available, constant-current temporary pacemaker programmed by the investigator to provide temporary pacing support. The StealthTrac Lead will remain inserted until the next calendar day, at a minimum, and will be removed once the clinical need for temporary pacing ends. The maximum duration of lead insertion is two (2) days following the lead insertion procedure.

Follow up evaluations will be performed for as long as the StealthTrac Lead remains inserted. Subjects will also undergo a 30-day post-removal follow-up before completing participation. On the final follow-up, prior to StealthTrac Lead removal, Subjects may be tested in multiple postures. Subjects with pacing capture in the upright posture may have ECGs recorded during various isometrics or while walking with pacing from the StealthTrac Lead.

Prior to removal, a final lead evaluation will be performed and fluoroscopy will be used to document the final lead position. Echocardiographic imaging will be obtained before and after the removal procedure to characterize any new or worsened pericardial effusions. A final post-removal follow-up will be performed in person or remotely to document any latent adverse events.

The overall study is expected to last four (4) months, comprising two (2) months for enrollment and follow-up and two (2) months to monitor study data and prepare a final report.

ELIGIBILITY:
Inclusion criteria

1. At least 18 years old
2. Subjects who:

   * Are undergoing one of the following planned (non-urgent) procedures that are associated with the potential need for temporary bradycardia pacing:

     * Transarterial transcatheter aortic valve implantation (TAVI)
     * Transarterial balloon aortic valvuloplasty (BAV)
     * Cardiovascular implantable electronic device (CIED) pulse generator replacement
     * Cardiovascular implantable electronic device (CIED) lead extraction OR
   * Subjects with bradycardia who are under evaluation to determine if the cause is transient or permanent

Exclusion criteria

1. BMI ≥ 35 kg/m2
2. Septic shock
3. Severe anemia
4. Patients on dual antiplatelet therapy or anti-coagulation that cannot be stopped for the procedure
5. Circumstances that prevent data collection or follow-up
6. Participation in any concurrent clinical study without prior written approval from the Sponsor
7. Inability or unwillingness to provide informed consent to participate in the Study

   Known prior history for any of the following:
8. Median or partial sternotomy
9. Acute coronary syndrome within past 90 days
10. NYHA Functional Classification IV within past 90 days
11. Surgically corrected congenital heart disease (not including catheter-based procedures)
12. Allergies to the device materials such as stainless steel, titanium, platinum, iridium, polyethylene, polyurethane, polycarbonate and silicone
13. Surgery with disruption of the lung, pericardium or connective tissue between the sternum and pericardium, including adhesions
14. Significant anatomic derangement of or within the thorax (e.g., pectus excavatum, significant scoliosis)
15. Thoracic radiation therapy, pneumothorax, pneumomediastinum or other medical treatments which may complicate the AtaCor EV Temporary Pacing Lead System insertion procedure
16. Any conditions which may complicate the AtaCor EV Temporary Pacing Lead System insertion procedure
17. Pericardial disease, pericarditis and mediastinitis
18. Medical treatments, surgeries or conditions that increase the potential for pericardial adhesions
19. FEV1 < 1 liter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-09-19 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-01-12 (Actual)

PRIMARY OUTCOMES:
Freedom from severe ADEs | Up to 30 days post-lead removal
  Freedom from Adverse Device Effects, CTCAE Grade 3 or Higher
Percentage of Subjects with pacing capture | Up to 2 days post-lead insertion
  Percentage of Subjects with demonstrated pacing capture following lead fixation

CONTACTS AND LOCATIONS:
Overall Officials: Martin C Burke, DO, Principal Investigator — AtaCor Medical, Inc.
Locations (1):
- University Hospital Center Split, Split, Croatia

IPD SHARING:
Plan to Share IPD: No